CLINICAL TRIAL: NCT03335514
Title: Changes of GALNT4 and the Relationship With PSGL-1on Monocytes and Hs-CRP in Blood of Patients With Coronary Heart Disease
Brief Title: GALNT4 in Patients With Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: LCKY2017
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Acute Coronary Syndrome
Keywords: GALNT4
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- STEMI: The study population consists of 20 patients with ST-elevated acute myocardial infarction (STEMI,n = 20) who are admitted within 24 hours after chest pain attack. They will all undergo coronary angiography. The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded.
  Interventions: Diagnostic Test: expression of GALNT4
- NSTE-ACS: The study population consists of 30 patients with non-ST elevated acute myocardial infarction (NSTE-ACS,n=30) who are admitted within 24 hours after chest pain attack. They will all undergo coronary angiography. The diagnosis is made according to American Heart Association (AHA, 2014 and 2015) guidelines. Patients who had autoimmune diseases, malignancies, chronic or acute infections, severe heart failure (NYHA class 3 and 4) and advanced liver or renal diseases are excluded.
  Interventions: Diagnostic Test: expression of GALNT4
- SAP: The study population consists of 30 patients with stable angina pectoris (SAP, n = 30). The diagnosis is made according to the criteria of the American Heart Association (AHA, 2014 and 2015). Patients who had autoimmune diseases, malignancies,chronic or acute infections, severe heart failure (NYHA class 3and 4) and advanced liver or renal diseases are excluded.
  Interventions: Diagnostic Test: expression of GALNT4
- CONTROL: 20 age and body mass index matched healthy subjects with neither coronary artery disease nor any of the components of the metabolic syndrome are studied as Normal group
  Interventions: Diagnostic Test: expression of GALNT4

INTERVENTIONS:
Diagnostic Test: expression of GALNT4 — Blood is obtained into ethylenediaminetetraacetic acid（EDTA） tubes from all subjects via antecubital venepuncture and the total RNA was extracted from blood.Realtime PCR was performed to measure the expression of GALNT4.

SUMMARY:
The expression of GALNT4 in blood with acute coronary syndrome

DETAILED DESCRIPTION:
Emerging evidences have linked GALNTs to cardiovascular disease or susceptibility to CAD.GALNT4, a member of the GalNAc-Ts family,contributes to the initiation of O-linked. Polymorphisms in GALNT4 have been linked with incidence of MI in an Irish population, probably that O-glycosylation of PSGL-1 by GalNAc-T4 may be important for many P-selectin mediated inflammation.However, there is few relevant studies about the expression of GALNT4 in patients with acute coronary syndrome.This study valuates the expression of GALNT4 in patients with acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as acute coronary syndrome,including STEMI,NSTE-ACS,or diagnosed as SAP by CAG.

  * with left ventricular ejection fraction（LVEF）>=45%
  * written informed consents are obtained
  * admitted within 24 hours after chest pain attacked(except SAP)

Exclusion Criteria:

* • complicated with rheumatic heart disease, coronary arteritis, hypertrophic cardiomyopathy or dilated cardiomyopathy

  * complicated with malignant tumor,the immune system diseases, blood system diseases, recently (within 2 weeks) taking glucocorticoid drugs, the use of immunosuppressive agents and cerebral infarction
  * with acute or chronic infection, surgery or trauma in the last month
  * secondary hypertension, severe liver dysfunction,severe renal insufficiency
  * with abnormal thyroid function or allergy to iodine agent
  * refusal to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALL the 4 groups will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
the expression of GALNT4 | 12 months
  Realtime RCR measure the expression of galnt4 in peripheral blood

SECONDARY OUTCOMES:
MACEs during 12-month follow-up | 12 months
  All major adverse cardiac events( MACEs) including death, myocardial infarction, heart failure are recorded

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Block H, Ley K, Zarbock A. Severe impairment of leukocyte recruitment in ppGalNAcT-1-deficient mice. J Immunol. 2012 Jun 1;188(11):5674-81. doi: 10.4049/jimmunol.1200392. Epub 2012 Apr 27. PMID 22544932
- [Background] Taylor DE. Plasmid-mediated tetracycline resistance in Campylobacter jejuni: expression in Escherichia coli and identification of homology with streptococcal class M determinant. J Bacteriol. 1986 Mar;165(3):1037-9. doi: 10.1128/jb.165.3.1037-1039.1986. PMID 3005233
- [Background] Beaman EM, Brooks SA. The extended ppGalNAc-T family and their functional involvement in the metastatic cascade. Histol Histopathol. 2014 Mar;29(3):293-304. doi: 10.14670/HH-29.293. Epub 2013 Oct 9. PMID 24105335
- [Background] Braenne I, Civelek M, Vilne B, Di Narzo A, Johnson AD, Zhao Y, Reiz B, Codoni V, Webb TR, Foroughi Asl H, Hamby SE, Zeng L, Tregouet DA, Hao K, Topol EJ, Schadt EE, Yang X, Samani NJ, Bjorkegren JL, Erdmann J, Schunkert H, Lusis AJ; Leducq Consortium CAD Genomicsdouble dagger. Prediction of Causal Candidate Genes in Coronary Artery Disease Loci. Arterioscler Thromb Vasc Biol. 2015 Oct;35(10):2207-17. doi: 10.1161/ATVBAHA.115.306108. Epub 2015 Aug 20. PMID 26293461
- [Background] O'Halloran AM, Patterson CC, Horan P, Maree A, Curtin R, Stanton A, McKeown PP, Shields DC. Genetic polymorphisms in platelet-related proteins and coronary artery disease: investigation of candidate genes, including N-acetylgalactosaminyltransferase 4 (GALNT4) and sulphotransferase 1A1/2 (SULT1A1/2). J Thromb Thrombolysis. 2009 Feb;27(2):175-84. doi: 10.1007/s11239-008-0196-z. Epub 2008 Feb 8. PMID 18259693